CLINICAL TRIAL: NCT02691949
Title: Efficacy and Safety of Mycophenolate Mofetil in subjectswithSjogren's Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Jeng-Hsien Yen, Professor, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S10418-4
Record Dates: First submitted 2016-02-16; First posted 2016-02-25 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mycophenolate mofetil standard (Experimental): mycophenolate mofetil 250mg 2# twice per day (BID)
  Interventions: Drug: Mycophenolate mofetil
- Mycophenolate sodium low (Experimental): mycophenolate mofetil 250mg 1# twice per day (BID)
  Interventions: Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Mycophenolate mofetil — mycophenolate mofetil 1# BID-2# BID

SUMMARY:
Past literature showed encouraging effects of mycophenolate on dryness symptoms and quality of life in patients with Sjogren's syndrome. Mycophenolate also has excellent immunomodulation effects in lupus nephritis. Currently Mycophenolate is only used in lupus nephritis and organ transplant. It is unknown whether low dosage of mycophenolate mofetil could be used to improve ocular dryness and oral dryness in patients with Sjogren's syndrome.

DETAILED DESCRIPTION:
Sjogren's syndrome is one of the most common autoimmune diseases in Taiwan. It is characterized by keratoconjunctivitis sicca and xerostomia. Although it is well established that Sjogren's syndrome is caused by infiltration and destruction of lacrimal gland and salivary gland by lymphocytic cells, effective treatment of patients' symptoms is lacking. Hydroxychloroquine is the most well-studied medication in Sjogren's syndrome. However, recent clinical trials showed disappointing effects of hydroxychloroquine in Sjogren's syndrome. Thus there is an unmet need to find effective treatment for patient's bothering symptoms.

Mycophenolate is a selective inhibitor of inosinemonophosphate dehydrogenase which leads to inhibition of the de novo pathway of nucleotide synthesis. The antiproliferative effect of mycophenolate mainly affects activated T and B lymphocytes because the proliferation of these cells is critically dependent on the de novo purine synthesis compared with other eukaryotic cells. Since these lymphocytes have been suggested to play a pivotal role in the inflammation and immunopathogenesis of Sjogren's syndrome, mycophenolate might be a promising agent in the treatment of Sjogren's syndrome.

Past literature showed encouraging effects of mycophenolate on dryness symptoms and quality of life in patients with Sjogren's syndrome. Mycophenolate also has excellent immunomodulation effects in lupus nephritis. Currently mycophenolate is only used in lupus nephritis and organ transplant. It is unknown whether low dosage of mycophenolate could be used to improve ocular dryness and oral dryness in patients with Sjogren's syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of primary Sjogren's syndrome based on the 2002 American-European Consensus criteria
2. Aged 20 to 75 years
3. Stable doses of oral corticosteroids(≦5mg/d) for at least 4 weeks before enrollment
4. Intolerance or inadequate response to hydroxychloroquine and (pilocarpine or cevimeline), defined as less than 50mm on at least 2 of VAS including:

   1. global assessment : 0mm (very bad) to 100mm (very good)
   2. pain: 0mm (very bad) to 100mm (very good)
   3. fatigue: 0mm (very bad) to 100mm (very good)
   4. xerostomia: 0mm (very bad) to 100mm (very good)
5. Adequate contraception for patients of childbearing potential

Exclusion Criteria:

1. Receiving biologics during the 6 previous months or any other immunosuppressant (methotrexate, cyclophosphamide, cyclosporine, azathioprine, mycophenolate mofetil (MMF), mycophenolate sodium, leflunomide, penicillamine) during the previous month
2. Any one of laboratory abnormalities:

   1. Serum creatinine ≥2 mg/dl
   2. aspartate aminotransferase (AST) or alanine transaminase (ALT) more than 1.5 x upper normal range of the laboratory
   3. Leukopenia (WBC<4000/μl)
   4. Hb ≤ 9 g/dl (5.6 mmol/l) for males and 8.5 g/dl (5.3 mmol/l) for females
   5. Neutrophil less than 1.5 x 109/l
   6. Platelet count less than 150 x 109/l
3. History of other autoimmune diseases
4. Use topical cyclosporine eyedrops, antihistamine, anticholinergic, antidepressant, or antipsychotic drug with possible effects on ocular dryness or oral dryness within 1 month
5. Pregnant or lactating women
6. Previous or current malignancies adequately controlled less than 5 years, hepatitis B, hepatitis C, HIV infection, tuberculosis, or diabetes
7. Subjects with serious infections requiring hospitalization within the last 12 months
8. Subjects with herpes zoster or cytomegalovirus that resolved less than 2 months before enrollment
9. Subjects who have received any live vaccines within 3 months
10. Underlying cardiac, pulmonary, metabolic, renal, hepatic, gastrointestinal, haematological or neurological conditions, chronic or latent infectious diseases or immune deficiency which places the patient at an unacceptable risk for participation in the study
11. History of recurring or chronic infections or underlying conditions which may further predispose patients to serious infection
12. Subjects who are impaired, incapacitated, or incapable of completing study-related assessments
13. History of allergy to mycophenolate sodium
14. Nausea, vomiting, diarrhea within 1 week before enrollment
15. History of psychosis, seizure, retinopathy
16. Infection 2 weeks before enrollment
17. Heart rate < 60/min at rest

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Change of Composite Index of Sjogren's syndrome | baseline, 28 week

SECONDARY OUTCOMES:
ocular dryness | baseline, 28 week
  We will calculate the change of ocular dryness from baseline to week 28 (0mm [very bad] to 100mm [very good])
physician visual analog scale (VAS) | baseline, 28 week
  We will calculate the change of physician VAS from baseline to week 28 (0mm [very bad] to 100mm [very good])
Schirmer's test | baseline, 28 week
  We will calculate the change of Schirmer's test results from baseline to week 28
Saxon's test | baseline, 28 week
  We will calculate the change of Saxon's test results from baseline to week 28
heart rate | baseline, 28 week
  resting heart rate
blood pressure | baseline, 28 week
  resting blood pressure
leukocyte count | baseline, 28 week
  WBC count
Hb level | baseline, 28 week
  Hb level
platelet count | baseline, 28 week
  platelet count

CONTACTS AND LOCATIONS:
Overall Officials: Jeng-Hsien Yen, Principal Investigator — Kaohsiung Medical University; Wen-Chan Tsai, Study Director — Kaohsiung Medical University; Tsan-Teng Ou, MD, Study Director — Kaohsiung Medical University; Cheng-Chin Wu, MD, Study Director — Kaohsiung Medical University; Wan-Yu Sung, MD, Study Director — Kaohsiung Medical University; Chia-Chun Tseng, MD, Study Director — Kaohsiung Medical University

IPD SHARING:
Plan to Share IPD: No
We won't share our data

REFERENCES:
- [Result] Willeke P, Schluter B, Becker H, Schotte H, Domschke W, Gaubitz M. Mycophenolate sodium treatment in patients with primary Sjogren syndrome: a pilot trial. Arthritis Res Ther. 2007;9(6):R115. doi: 10.1186/ar2322. PMID 17986340